CLINICAL TRIAL: NCT03713619
Title: A Randomized, Double-blind, Multi-center Study Assessing Short (16 Weeks) and Long-term Efficacy (up to 1 Year), Safety, and Tolerability of 2 Subcutaneous Secukinumab Dose Regimens in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (SUNSHINE).
Brief Title: This Was a Study of Efficacy and Safety of Two Secukinumab Dose Regimens in Subjects With Moderate to Severe Hidradenitis Suppurativa (HS).
Acronym: SUNSHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457M2301; 2018-002063-26 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: acne inversa; Hidradenitis suppurativa; maladie de Verneuil; inflammatory disease; AIN457; AIN457M; secukinumab; HS; lumps; skin; lesions
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This was a Multicenter, randomized, double-blind, placebo-controlled, parallel group study, with two secukinumab dose regimens in 541 patients with moderate to severe HS.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- secukinumab 1 (Active Comparator): Secukinumab 300mg every 2 weeks
  Interventions: Drug: secukinumab
- secukinumab 2 (Active Comparator): Secukinumab 300mg every 4 weeks
  Interventions: Drug: secukinumab
- placebo 1 (Placebo Comparator): Placebo group to secukinumab 300mg every 2 weeks
  Interventions: Drug: Placebo
- placebo 2 (Placebo Comparator): Placebo group to secukinumab 300mg every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: secukinumab — Secukinumab 300mg every 2 or every 4 weeks
  Other Names: AIN457
  Arms: secukinumab 1; secukinumab 2
Drug: Placebo — Placebo 300mg every 2 or every 4 weeks
  Arms: placebo 1; placebo 2

SUMMARY:
The purpose of this study was to demonstrate superiority of secukinumab at Week 16, based on Hidradenitis Suppurativa Clinical Response (HiSCR) rates versus placebo, along with the maintenance of efficacy of secukinumab at Week 52 in subjects with moderate to severe HS. Moreover, this study also assessed the safety and tolerability of secukinumab.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled, parallel group study with two secukinumab dose regimens in 541 patients with moderate to severe HS. The study consisted of: screening (up to 4 weeks) treatment period 1 (16 weeks, active drug or placebo) and treatment period 2 (up to 1 year all patients on active drug); there was an optional extension study (NCT04179175). Adult males and females with moderate to severe HS were included, with a diagnosis of HS greater than 1 year prior to baseline. Dosing was once every 2 weeks, or once every 4 weeks via pre-filled syringe; periodic home-dosing is included.

In Treatment Period 1, participants were randomized to secukinumab Q2W, secukinumab Q4W, placebo Q2W or placebo Q4W in 1:1:0.5:0.5 ratio. In Treatment Period 2, at the Week 16 visit participants initially randomized to placebo were switched to one of the two active dose regimens (secukinumab Q2W or Q4W), while subjects randomized to secukinumab during Treatment Period 1 continued on the same dose.

At the Week 16 visit, subjects initially randomized to placebo were switched to one of the two active dose regimens (secukinumab Q2W or Q4W), while subjects randomized to secukinumab during Treatment Period 1 continued on the same dose.

The primary objective was to demonstrate the efficacy of secukinumab compared to placebo with respect to HISCR after 16 weeks of treatment; secondary objectives were to assess difference in proportion of patients with HS flares, and proportion of patients with clinical response in HS related skin pain after 16 weeks of treatment. Key safety data was collected, along with Patient Reported Outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female patients ≥ 18 years of age.
* Diagnosis of HS ≥ 1 year prior to baseline.
* Patients with moderate to severe HS defined as:
* A total of at least 5 inflammatory lesions, i.e. abscesses and/or inflammatory nodules AND
* Inflammatory lesions should affect at least 2 distinct anatomic areas
* Patients agree to daily use of topical over-the-counter antiseptics on the areas affected by HS lesions while on study treatment.

Exclusion Criteria:

* Total fistulae count ≥ 20 at baseline.
* Any other active skin disease or condition that may interfere with assessment of HS.
* Active ongoing inflammatory diseases other than HS that require treatment with prohibited medications.
* Use or planned use of prohibited treatment. Washout periods detailed in the protocol have to be adhered to.
* History of hypersensitivity to any of the study drug constituents.
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (108):
- United States (18):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Rogers, Arkansas
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Glenview, Illinois
  - Novartis Investigative Site, West Dundee, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New Brighton, Minnesota
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Fairborn, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Argentina (3):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Phillip, Australian Capital Territory
  - Novartis Investigative Site, Benowa, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Brussels, Brussels Capital, Belgium
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
- Czechia (2):
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Pilsen
- France (8):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (8):
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Potsdam
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
- India (4):
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (4):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Nakagami, Okinawa
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
- Philippines (3):
  - Novartis Investigative Site, Davao City, Davao Region
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Las Piñas
- Poland (3):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Ossy
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Slovakia (2):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Martin
- Novartis Investigative Site, Seoul, South Korea
- Spain (6):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
- Novartis Investigative Site, Uppsala, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Gaziantep
- United Kingdom (6):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Barnsley
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Alavi A, Reguiai Z, Jemec GBE, Gottlieb AB, Wozniak MB, Uhlmann L, Fan H, Llobet Martinez A, Bruin G, Thomas N, Alarcon I, Bieth B, Ravichandran S, Kimball AB. Secukinumab in the Treatment of Moderate-to-Severe Hidradenitis Suppurativa: Pooled Pharmacokinetics and Safety Results From the SUNSHINE and SUNRISE Phase 3 Studies. Int J Dermatol. 2026 Feb;65(2):289-298. doi: 10.1111/ijd.70025. Epub 2025 Aug 21. PMID 40839197
- [Derived] Ingram JR, Szepietowski JC, Matusiak L, Kokolakis G, Wozniak MB, Ortmann CE, Martinez AL, Ravichandran S, Thomas N, Alarcon I, Pieterse CC, Alam MS, Ioannides D, Kimball AB. Assessing Long-Term Pain Reduction with Secukinumab in Moderate to Severe Hidradenitis Suppurativa: A Post Hoc Analysis of the SUNSHINE and SUNRISE Phase 3 Trials. Dermatol Ther (Heidelb). 2025 Jul;15(7):1833-1849. doi: 10.1007/s13555-025-01426-x. Epub 2025 May 15. PMID 40372667
- [Derived] Zouboulis CC, Kyrgidis A, Alavi A, Jemec GBE, Martorell A, Marzano AV, van der Zee HH, Wozniak MB, Martinez AL, Kasparek T, Bachhuber T, Ortmann CE, Lobach I, Thomas N, Ravichandran S, Tzellos T. Secukinumab efficacy in patients with hidradenitis suppurativa assessed by the International Hidradenitis Suppurativa Severity Score System (IHS4): A post hoc analysis of the SUNSHINE and SUNRISE trials. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1421-1430. doi: 10.1111/jdv.20369. Epub 2024 Oct 19. PMID 39425517
- [Derived] Passera A, Muscianisi E, Demanse D, Okoye GA, Jemec GBE, Mayo T, Hsiao J, Shi VY, Byrd AS, Wei X, Uhlmann L, Vandemeulebroecke M, Ravichandran S, Porter ML. New insights on hidradenitis suppurativa phenotypes and treatment response: An exploratory automated analysis of the SUNSHINE and SUNRISE trials. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1410-1420. doi: 10.1111/jdv.20234. Epub 2024 Aug 5. PMID 39101698
- [Derived] Kimball AB, Jemec GBE, Alavi A, Reguiai Z, Gottlieb AB, Bechara FG, Paul C, Giamarellos Bourboulis EJ, Villani AP, Schwinn A, Rueff F, Pillay Ramaya L, Reich A, Lobo I, Sinclair R, Passeron T, Martorell A, Mendes-Bastos P, Kokolakis G, Becherel PA, Wozniak MB, Martinez AL, Wei X, Uhlmann L, Passera A, Keefe D, Martin R, Field C, Chen L, Vandemeulebroecke M, Ravichandran S, Muscianisi E. Secukinumab in moderate-to-severe hidradenitis suppurativa (SUNSHINE and SUNRISE): week 16 and week 52 results of two identical, multicentre, randomised, placebo-controlled, double-blind phase 3 trials. Lancet. 2023 Mar 4;401(10378):747-761. doi: 10.1016/S0140-6736(23)00022-3. Epub 2023 Feb 3. PMID 36746171
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1839

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in 111 study sites worldwide.
Groups:
- Secukinumab - Q2W: Secukinumab 300mg every 2 weeks (Treatment Period 1 and 2)
- Secukinumab - Q4W: Secukinumab 300mg every 4 weeks (Treatment Period 1 and 2)
- Placebo: Placebo group to secukinumab 300mg (Treatment Period 1)
- Placebo - Re-randomized to Secukinumab Q2W: Placebo group, re-randomized to secukinumab 300mg Q2W at week 16 (Treatment Period 2)
- Placebo - Re-randomized to Secukinumab Q4W: Placebo group, re-randomized to secukinumab 300mg Q4W at week 16 (Treatment Period 2)
Period: Treatment Period 1 (Until Week 16)
Arm/Group | Secukinumab - Q2W | Secukinumab - Q4W | Placebo | Placebo - Re-randomized to Secukinumab Q2W | Placebo - Re-randomized to Secukinumab Q4W
Started | 182 | 181 | 181 | 0 | 0
Full Analysis Set (FAS) (The FAS excluded participants who were misrandomized or had severe GCP violations) | 181 | 180 | 180 | 0 | 0
Completed | 168 | 169 | 172 | 0 | 0
Not Completed | 14 | 12 | 9 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 0 | 0
Not completed — Technical problems | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 9 | 5 | 0 | 0
Not completed — Misrandomized | 0 | 0 | 1 | 0 | 0
Not completed — Severe GCP Violation | 1 | 1 | 0 | 0 | 0
Period: Treatment Period 2 (After Week 16)
Arm/Group | Secukinumab - Q2W | Secukinumab - Q4W | Placebo | Placebo - Re-randomized to Secukinumab Q2W | Placebo - Re-randomized to Secukinumab Q4W
Started | 168 | 169 | 0 | 85 | 87
Completed | 131 | 137 | 0 | 68 | 75
Not Completed | 37 | 32 | 0 | 17 | 12
Not completed — Adverse Event | 6 | 5 | 0 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 26 | 20 | 0 | 10 | 6
Not completed — Poor efficacy | 1 | 2 | 0 | 2 | 1
Not completed — Lost to Follow-up | 3 | 3 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Secukinumab 1 - Q2W: Secukinumab 300mg every 2 weeks
- Secukinumab 2 - Q4W: Secukinumab 300mg every 4 weeks
- Placebo: Placebo group to secukinumab 300mg every 4 weeks
- Total: Total of all reporting groups
Arm/Group | Secukinumab 1 - Q2W | Secukinumab 2 - Q4W | Placebo | Total
Number analyzed (Participants) | 181 | 180 | 180 | 541
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 178 | 177 | 179 | 534
  >=65 years | 3 | 3 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.53) | 35.7 (11.71) | 35.5 (10.75) | 36.1 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 100 | 102 | 304
  Male | 79 | 80 | 78 | 237
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 145 | 146 | 139 | 430
  Black or African American | 15 | 10 | 12 | 37
  Asian | 19 | 23 | 24 | 66
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Multiple | 1 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hidradenitis Suppurativa Clinical Response (HiSCR50)
Description: HiSCR50 at Week 16 is defined as at least a 50% decrease in Abscess and inflammatory Nodule (AN) count compared to baseline with no increase in the number of abscesses and/or in the number of draining fistulas from baseline to Week 16. The baseline is defined as the last assessment (including unscheduled visits) obtained before/on the day of the first administration of the study treatment, or on the randomization date if there had been no drug administration.
  This endpoint was analyzed by logistic regression.
Time Frame: 16 weeks
Population: Full analysis set (FAS)
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Placebo group to secukinumab 300mg
Arm/Group | Secukinumab 1 - Q2W | Secukinumab 2 - Q4W | Placebo
Number analyzed (Participants) | 181 | 180 | 180
Percentage of participants | 45.0 | 41.8 | 33.7
Statistical Analysis 1: Comparison: Secukinumab 1 - Q2W vs Placebo; Logistic regression analysis of HiSCR50 response at Week 16 (multiple imputation); Test type: Superiority; p = 0.0070, Regression, Logistic; Odds Ratio, log = 1.75, 95% CI 2-sided [1.12 to 2.73]
Statistical Analysis 2: Comparison: Secukinumab 2 - Q4W vs Placebo; Logistic regression analysis of HiSCR50 response at Week 16 (multiple imputation); Test type: Superiority; p = 0.0418, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.95 to 2.32]

2. Secondary Outcome: Percentage Change From Baseline in AN50 Count at Week 16
Description: The HS affected areas, e.g. right and left axillary (armpit), right and left gluteal ("buttock"), right and left inguinal-femoral (groin), perineal, pubic, sternal, right and left sub-mammary (breast) and others were assessed by the physician for abscesses, inflammatory nodules, draining fistulas, total fistulas, and other lesions.
  Inflammatory lesions, including abscesses, nodules, draining fistulae, total fistulae and other lesions were counted. The analysis method for percentage change from baseline in abscesses and inflammatory nodules (AN) count at Week 16 was an ANCOVA model.
Time Frame: Baseline, 16 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Secukinumab 1 - Q2W | Secukinumab 2 - Q4W | Placebo
Number analyzed (Participants) | 181 | 180 | 180
percentage change from baseline | -46.8 (3.33) | -42.4 (4.01) | -24.3 (4.33)
Statistical Analysis 1: Comparison: Secukinumab 1 - Q2W vs Placebo; Analysis of covariance of percentage change from baseline in AN count at Week 16 (multiple imputation); Test type: Superiority; p < 0.0001, ANCOVA; Least square Mean Difference = -23.05, 95% CI 2-sided [-33.90 to -12.21]
Statistical Analysis 2: Comparison: Secukinumab 2 - Q4W vs Placebo; Analysis of covariance of percentage change from baseline in AN count at Week 16 (multiple imputation); Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean difference = -18.46, 95% CI 2-sided [-29.32 to -7.60]

3. Secondary Outcome: Percentage of Participants With Hidradenitis Suppurativa (HS) Flares
Description: Percentage of participants who experience at least one flare over 16 weeks. A flare is defined as at least a 25% increase in abscesses and inflammatory nodules (AN) count with a minimum increase of 2 AN relative to baseline.
  This endpoint was analyzed by logistic regression.
Time Frame: 16 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Groups:
- Placebo 2: Placebo group to secukinumab 300mg
Arm/Group | Secukinumab 1 - Q2W | Secukinumab 2 - Q4W | Placebo 2
Number analyzed (Participants) | 181 | 180 | 180
Percentage of participants | 15.4 | 23.2 | 29.0
Statistical Analysis 1: Comparison: Secukinumab 1 - Q2W vs Placebo 2; Logistic regression analysis of Flare over 16 weeks (multiple imputation); Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio, log = 0.42, 95% CI 2-sided [0.25 to 0.73]
Statistical Analysis 2: Comparison: Secukinumab 2 - Q4W vs Placebo 2; Logistic regression analysis of Flare over 16 weeks (multiple imputation); Test type: Superiority; p = 0.0926, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.43 to 1.17]

4. Secondary Outcome: Percentage of Participants Achieving NRS30
Description: Patients achieving Numerical Rating Scale score of 30 (NRS30) at week 16, defined as at least a 30% reduction and at least one unit reduction from baseline in the Patient's Global assessment of Skin Pain (where range 0 [no skin pain] to 10 [worst skin pain]).
  This endpoint was analyzed by logistic regression.
Time Frame: Baseline, week 16
Population: FAS restricted to participants with baseline NRS score greater or equal to 3
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 1 - Q2W | Secukinumab 2 - Q4W | Placebo
Number analyzed (Participants) | 131 | 123 | 119
Percentage of participants | 34.1 | 32.2 | 23.8
Statistical Analysis 1: Comparison: Secukinumab 1 - Q2W vs Placebo; Logistic regression analysis of skin pain/NRS30 response at Week 16 (pooled data, multiple imputation); Test type: Superiority; p = 0.0248, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.00 to 3.40]
Statistical Analysis 2: Comparison: Secukinumab 2 - Q4W vs Placebo; Logistic regression analysis of skin pain/NRS30 response at Week 16 (pooled data, multiple imputation); Test type: Superiority; p = 0.0044, Regression, Logistic; Odds Ratio, log = 1.77, 95% CI 2-sided [1.15 to 2.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from first dose of study treatment, up to approximately 60 weeks for AIN457 (up to 52 weeks for subjects moving to extension study) and 16 weeks for placebo.
Description: AEs are any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Groups:
- AIN457 Q2W: Subjects who were randomized to AIN457 (secukinumab) 300mg Q2W dose regimen at the study entry. Adverse events were assessed up to Week 60
- AIN457 Q4W: Subjects who were randomized to AIN457 (secukinumab) 300mg Q4W dose regimen at the study entry. Adverse events were assessed up to Week 60
- Placebo: Subjects received matching placebo up to 16 weeks
- Any AIN457 Q2W: Subjects who received at least 1 dose of secukinumab 300 mg Q2W dose (e.g., subjects who switched from placebo to secukinumab Q2W at Week 16). Adverse events were assessed up to Week 60
- Any AIN457 Q4W: Subjects who received at least 1 dose of secukinumab 300 mg Q4W dose (e.g., subjects who switched from placebo to secukinumab Q4W at Week 16). Adverse events were assessed up to Week 60
- Any AIN457: Subjects who received at least 1 dose of secukinumab
Arm/Group | AIN457 Q2W | AIN457 Q4W | Placebo | Any AIN457 Q2W | Any AIN457 Q4W | Any AIN457
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/180 | 0/180 | 0/266 | 0/267 | 0/533
Serious Adverse Events (participants affected / at risk) | 13/181 | 9/180 | 6/180 | 18/266 | 19/267 | 37/533
Other Adverse Events (participants affected / at risk) | 135/181 | 132/180 | 88/180 | 184/266 | 183/267 | 367/533
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2W (N=181) | AIN457 Q4W (N=180) | Placebo (N=180) | Any AIN457 Q2W (N=266) | Any AIN457 Q4W (N=267) | Any AIN457 (N=533)
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2
Breast cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Large intestine infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sweat gland infection (Infections and infestations) | 1 | 3 | 0 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1
C3 glomerulopathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 4 | 4 | 8
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2W (N=181) | AIN457 Q4W (N=180) | Placebo (N=180) | Any AIN457 Q2W (N=266) | Any AIN457 Q4W (N=267) | Any AIN457 (N=533)
Abdominal pain (Gastrointestinal disorders) | 7 | 6 | 1 | 8 | 10 | 18
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 1 | 4 | 9 | 13
Constipation (Gastrointestinal disorders) | 1 | 5 | 0 | 1 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 11 | 16 | 9 | 12 | 24 | 36
Nausea (Gastrointestinal disorders) | 4 | 8 | 7 | 6 | 13 | 19
Toothache (Gastrointestinal disorders) | 7 | 6 | 4 | 9 | 7 | 16
Vomiting (Gastrointestinal disorders) | 5 | 7 | 0 | 6 | 9 | 15
Asthenia (General disorders) | 3 | 4 | 4 | 5 | 4 | 9
Chest pain (General disorders) | 0 | 5 | 0 | 0 | 5 | 5
Fatigue (General disorders) | 6 | 11 | 8 | 8 | 13 | 21
Pyrexia (General disorders) | 13 | 8 | 2 | 16 | 12 | 28
Hepatic steatosis (Hepatobiliary disorders) | 4 | 2 | 2 | 4 | 3 | 7
Bronchitis (Infections and infestations) | 5 | 6 | 3 | 5 | 8 | 13
COVID-19 (Infections and infestations) | 5 | 3 | 0 | 6 | 7 | 13
Cellulitis (Infections and infestations) | 4 | 3 | 4 | 6 | 6 | 12
Conjunctivitis (Infections and infestations) | 5 | 4 | 1 | 5 | 6 | 11
Ear infection (Infections and infestations) | 3 | 4 | 0 | 3 | 4 | 7
Folliculitis (Infections and infestations) | 4 | 4 | 2 | 6 | 4 | 10
Fungal skin infection (Infections and infestations) | 4 | 0 | 0 | 4 | 0 | 4
Gastroenteritis (Infections and infestations) | 8 | 4 | 1 | 8 | 4 | 12
Influenza (Infections and infestations) | 1 | 6 | 4 | 1 | 6 | 7
Nasopharyngitis (Infections and infestations) | 32 | 24 | 13 | 40 | 29 | 69
Pharyngitis (Infections and infestations) | 7 | 5 | 1 | 8 | 7 | 15
Sinusitis (Infections and infestations) | 4 | 2 | 2 | 7 | 2 | 9
Suspected COVID-19 (Infections and infestations) | 5 | 3 | 0 | 6 | 7 | 13
Tonsillitis (Infections and infestations) | 6 | 2 | 1 | 7 | 4 | 11
Upper respiratory tract infection (Infections and infestations) | 9 | 13 | 4 | 12 | 17 | 29
Urinary tract infection (Infections and infestations) | 9 | 8 | 3 | 10 | 10 | 20
Vulvovaginal candidiasis (Infections and infestations) | 4 | 2 | 0 | 4 | 3 | 7
Vulvovaginal mycotic infection (Infections and infestations) | 6 | 2 | 1 | 7 | 4 | 11
Ligament sprain (Injury, poisoning and procedural complications) | 6 | 4 | 0 | 8 | 4 | 12
Amylase increased (Investigations) | 3 | 4 | 0 | 3 | 5 | 8
Lipase increased (Investigations) | 8 | 7 | 2 | 8 | 9 | 17
SARS-CoV-2 test negative (Investigations) | 6 | 5 | 2 | 8 | 7 | 15
SARS-CoV-2 test positive (Investigations) | 2 | 4 | 0 | 4 | 5 | 9
Weight increased (Investigations) | 2 | 5 | 2 | 3 | 5 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 4 | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 8 | 14 | 9 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 8 | 7 | 12 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5 | 5 | 5 | 10
Dizziness (Nervous system disorders) | 6 | 3 | 3 | 7 | 5 | 12
Headache (Nervous system disorders) | 33 | 32 | 14 | 39 | 46 | 85
Migraine (Nervous system disorders) | 5 | 1 | 0 | 5 | 3 | 8
Depression (Psychiatric disorders) | 4 | 2 | 2 | 6 | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 1 | 7 | 10 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 3 | 11 | 7 | 18
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 2 | 9 | 4 | 13
Acne (Skin and subcutaneous tissue disorders) | 4 | 5 | 2 | 5 | 6 | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 4 | 5 | 9
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 3 | 6 | 9
Eczema (Skin and subcutaneous tissue disorders) | 8 | 6 | 1 | 9 | 9 | 18
Hidradenitis (Skin and subcutaneous tissue disorders) | 16 | 17 | 23 | 28 | 26 | 54
Intertrigo (Skin and subcutaneous tissue disorders) | 10 | 7 | 2 | 11 | 8 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 6 | 2 | 15 | 8 | 23
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 5 | 1 | 6 | 5 | 11
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 6 | 5 | 11
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 4 | 5 | 2 | 6 | 6 | 12
Hypertension (Vascular disorders) | 6 | 4 | 2 | 8 | 5 | 13
White blood cell count increased (Investigations) | 1 | 2 | 4 | 3 | 2 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 4 | 2 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03713619/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03713619/SAP_001.pdf